CLINICAL TRIAL: NCT01610375
Title: Telephone Follow-up After Treatment for Endometrial Cancer.
Acronym: TEACUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TEACUP
Record Dates: First submitted 2012-03-22; First posted 2012-06-04 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telephone Follow-up (Other): Women previously treated for endometrial cancer will be recruited into one study group and continue to be followed per the current routine clinic follow-up. However, an additional program (telephone follow-up) will be offered in parallel to the current clinic follow-up. Outcomes obtained from the telephone follow-up will be compared with the current clinical assessment.
  Interventions: Other: Telephone Follow-up

INTERVENTIONS:
Other: Telephone Follow-up — This is a non-randomised observational study to assess the value of a symptom checklist to detect recurrence in women with endometrial cancer. Women will be telephoned using an evidence-based symptom checklist in parallel to the standard clinic-based follow-up. The researcher will call the participants 2 to 5 days prior to their scheduled clinic review dates to enquire about the presence of symptoms which may be indicative of disease recurrence. In addition, the researcher will also enquire about the participants' wellbeing and provide standard lifestyle resource on physical activity, diet and other lifestyle behaviours and supportive care when needed.
  Other Names: TEACUP

SUMMARY:
The aim of this study is to investigate the feasibility, safety and accuracy of a telephone follow-up for women previously treatment for endometrial cancer.

To achieve this aim, potentially eligible women attending the Queensland Centre for Gynaecological Cancer (QCGC) outpatient clinic for review following previous treatment for endometrial cancer will be recruited by this study. The study aims to recruit all new patients as well as all patients who return to QCGC for their follow-up and who had treatment within the previous 2 years.

The proposed project will involve generation of an evidence-based checklist of signs and symptoms of disease recurrence from a thorough literature review. The generated symptom checklist will be pilot tested and the refined symptom checklist will be used to follow study participants over a period of 12 months.

During the follow-up period, the basic standard of follow-up after primary treatment for endometrial cancer at the QCGC, Royal Brisbane and Women's Hospital (RBWH)will not be altered; however, the study participants will be interview via telephone 2 to 5 days prior to their scheduled review dates.

The main outcome measure will be the estimated recurrence rate as derived from the telephone assessment and this will be compared to the clinically detected recurrences as recorded in patients' medical files.

It is hypothesized, that the telephone follow-up will identify 90% of all recurrences correctly that are later confirmed during the clinical follow-up.

In addition to the main outcome, we will also assess patients' satisfaction with each of the follow-up programs, whether or not lifestyle behaviours were queried and support offered to improve wellbeing.

DETAILED DESCRIPTION:
The focus of the study is;

1. To generate an evidence-based checklist of signs and symptoms of recurrence of endometrial cancer.
2. To assess the sensitivity and specificity of a telephone follow-up compared to the current clinic-based follow-up in the detection of recurrence of endometrial cancer.
3. To determine patients' satisfaction with the clinic and telephone follow-up.
4. To assess patients' self reported well being (physical activity, smoking, diet, anxiety, depression and quality of life).

The proposed project will involve generation of an evidence-based checklist of signs and symptoms of recurrence. The generated symptom checklist will be used to follow study participants over a period of 12 months.

During the follow-up period, patients' routine clinic follow-up schedules will not be altered, however; the study participants will be interviewed via telephone 2 to 5 days prior to their scheduled clinic visits dates. The checklist of signs and symptoms generated by this study will form the basis for this interview.

In addition, we will also enquire about the participant's wellbeing and provide resources on physical activity, diet and other life style behaviours and supportive care when needed.

The data analysis will include determining:

i. Sensitivity- Proportion of those with the condition who have a positive test.

ii. Specificity-Proportion of those without the condition who have a negative test.

iii. Positive predictive value (PV+) - Proportion of those with a positive test who have the condition.

iv. Negative predictive value (PV-) - Proportion of those with a negative test who do not have the condition.

Overall accuracy of the symptom checklist compared to the clinic-based follow-up program will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this pilot study, the patient must;

* Have completed primary treatment for endometrial cancer
* Be recurrence-free
* In the first to third year after treatment
* Be able to read and understand English
* Must have access to a telephone and adequate hearing
* Participants must be willing to complete questionnaire on satisfaction with nurse and clinic follow-up

Exclusion Criteria:

* Patients with disease recurrent or relapse
* Patients with metastatic disease presentation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity and overall accuracy of the telephone follow-up compared to clinic-based follow-up and patients' satisfaction. | 12 months
  The proposed project will involve generation of an evidence-based checklist of signs and symptoms of recurrence from a thorough literature review. The generated symptom checklist will be pilot tested and used in a one year prospective cohort study.

SECONDARY OUTCOMES:
Changes in lifestyle behaviours and quality of life overtime. | 12 months
  The researcher will conduct a telephone interview and will enquire about the participant's wellbeing and provide resources on physical activity, quality of life, diet, anxiety and depression and supportive care when needed prior to each clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, MD FRANZCOG CGO, Study Chair — Queensland Center for Gynecological Cancer; Monika Janda, PhD, Study Director — Queensland University of Technology
Locations (1):
- Royal Brisbane and Women's Hospital, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No